CLINICAL TRIAL: NCT00329797
Title: A Phase III Randomized Study to Evaluate the Efficacy of Zometa® for the Prevention of Osteoporosis and Associated Fractures in Patients Receiving Radiation Therapy and Long Term LHRH Agonists for High-Grade and/or Locally Advanced Prostate Cancer
Brief Title: Zoledronate in Preventing Osteoporosis and Bone Fractures in Patients With Locally Advanced Nonmetastatic Prostate Cancer Undergoing Radiation Therapy and Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG 0518; CDR0000476469; NCI-2009-00884 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Osteoporosis; Prostate Cancer
Keywords: osteoporosis; adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms | interventions — Calcium; Zoledronic Acid; Radiotherapy; Gonadotropin-Releasing Hormone; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic Acid (Experimental): Zoledronic acid q 6 months plus Vitamin D and calcium supplement for 3 years in addition to concurrent radiation therapy and LHRH therapy.
  Interventions: Dietary Supplement: Calcium; Dietary Supplement: Zoledronic acid; Radiation: radiation therapy; Drug: LHRH; Dietary Supplement: Vitamin D
- Control (Active Comparator): Vitamin D and calcium supplement everyday for 3 years in addition to concurrent radiation therapy and LHRH therapy.
  Interventions: Dietary Supplement: Calcium; Radiation: radiation therapy; Drug: LHRH; Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Calcium — A single dose of 500 mg of elemental calcium orally each day for 3 years.
Dietary Supplement: Zoledronic acid — Patients receive IV over 15 minutes once every 6 months for 3 years. The goal dose of zoledronic acid is 4 mg, but the selection of dose is determined based on calculated creatinine clearance at baseline.
  Other Names: Zometa; zoledronate
  Arms: Zoledronic Acid
Radiation: radiation therapy — Patients must receive external beam irradiation, brachytherapy (HDR or LDR), or a combination of external beam irradiation and brachytherapy at the discretion of the treating physician. Dose/duration also will be at the discretion of the treating physician; however, dose will not exceed 45 Gy to 100% of the proximal femur, and no proximal femur will receive ≥ 60 Gy.
Drug: LHRH — LHRH therapy must take place for a minimum of one year. Choice of LHRH agonist, dose, and duration are at the discretion of the treating physician.
Dietary Supplement: Vitamin D — 400 IU (10μg), orally each day for 3 years.

SUMMARY:
RATIONALE: Zoledronate may prevent bone loss in patients with prostate cancer undergoing radiation therapy and hormone therapy. It is not yet known whether zoledronate is more effective than calcium and vitamin D alone in preventing osteoporosis and bone fractures in patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying zoledronate to see how well it works compared to calcium and vitamin D alone in preventing osteoporosis and bone fractures in patients with locally advanced nonmetastatic prostate cancer undergoing radiation therapy and hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the potential benefit of bisphosphonate therapy comprising zoledronate plus vitamin D and calcium supplement vs standard therapy with vitamin D and calcium supplement in the prevention of osteoporosis and associated bone fractures in patients with locally advanced nonmetastatic adenocarcinoma of the prostate undergoing radiotherapy and luteinizing hormone-releasing hormone (LHRH) agonist therapy.

Secondary

* Evaluate the potential benefit of these regimens on quality of life in these patients.
* Evaluate the potential benefit in bone mineral density over a period of 3 years for patients treated with these regimens.

OUTLINE: This is randomized multicenter study. Patients are stratified according to T score of the hip by dual x-ray absorptiometry (DXA) scan (< -1.0 but > -2.5 vs ≥ - 1.0) and planned duration of luteinizing hormone-releasing hormone (LHRH) agonist therapy (1-2½ years vs > 2½ years). Patients are randomized to 1 of 2 treatment arms.

Quality of life is assessed at baseline and every 6 months during treatment.

ELIGIBILITY:
Eligibility criteria:

* Pathologically (histologically or cytologically) proven diagnosis of adenocarcinoma of the prostate within 12 months of registration;
* Any one of the following clinical stages:

  * T3 disease, any N stage, M0 with any Gleason score and any prostate-specific antigen (PSA); < T3 stage, any N stage, M0 with Gleason's score ≥ 8 and any PSA; < T3 stage, any N stage, M0 with Gleason's score 7 and PSA ≥ 15 nanograms/ml; < T3 stage, any N stage, M0 with Gleason score < 7 and PSA ≥ 20 nanograms/ml.
* A negative bone scan for metastatic disease;
* It is mandatory that the treating physician determine the planned duration of LHRH therapy prior to the site registering the patient (minimum 1 year of therapy); If patient is receiving pre-treatment LHRH therapy, it must have begun ≤ 6 months prior to registration. If pelvic radiation therapy (RT) has started, it must have begun ≤ 8 weeks prior to registration;
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup to be done within 16 weeks prior to registration:
* History/physical examination;
* Dental evaluation, including history of dental surgery (e.g., extraction or implant);
* Bone scan;
* T and L spine films;
* DXA scan: To be eligible the patient must have a scan on Lunar, Hologic, or Norland equipment only and the T scores in both the L spine and total hip must be > negative 2.5;
* Zubrod Performance Status 0-1 within 16 weeks prior to registration; (8/16/07)
* Age ≥ 18;
* Serum creatinine within 4 weeks prior to registration (8/16/07)
* Corrected serum calcium ≥ 8.4 and ≤ 10.6 mg/dl within 8 weeks prior to registration; note: for patients with an albumin of 4.0, corrected calcium=measured calcium. The formula for corrected calcium if serum albumin value is above or below 4.0 is as follows: Corrected calcium (mg/dl) = (4 - [patient's albumin (g/dl)] x 0.8) + patient's measured calcium (mg/dl)
* Patients who are sexually active must be willing/able to use medically acceptable forms of contraception, as the treatment involved in this study may be significantly teratogenic.
* Patient agrees to refrain from using all products listed in Section 9.2, "Non-permitted Supportive Therapy";
* Post-prostatectomy patients are eligible.
* Patient must sign study specific informed consent prior to study entry.

Ineligibility criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; e.g., carcinoma in situ of the breast or oral cavity are permissible;
* Patients with baseline T scores of ≤ -2.5 are excluded.
* Patients with baseline calculated creatinine clearance < 30 mL/min (estimated by Cockcroft-Gault formula below) are excluded. creatinine clearance male = [(140 - age) x (wt in kg)] / [(serum creatinine) x (72)]
* Prior bisphosphonate therapy;
* Prior pelvic radiation (other than for current prostate cancer) or prior systemic radiotherapeutic agents, such as strontium or samarium;
* Patients receiving systemic chemotherapy, steroids, growth hormones, or calcitonin;
* Patients with a history of Paget's disease or with uncontrolled thyroid or parathyroid dysfunction or with other diseases that influence bone metabolism;
* Known hypersensitivity to zoledronic acid or other bisphosphonates;
* Active dental problems at study entry, including infection of the teeth or jawbone; dental or fixture trauma; or a current or prior diagnosis of osteonecrosis of the jaw, exposed bone in the mouth, or slow healing after dental procedures;
* Recent or planned

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A. Lawton, MD, Principal Investigator — Medical College of Wisconsin; Matthew R. Smith, MD, Study Chair — Massachusetts General Hospital; Margaret Chamberlain-Wilmoth, PhD, MSS, RN, Study Chair — Carolinas Medical Center - University
Locations (88):
- United States (80):
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Lourdes Regional Cancer Center, Binghamton, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
- Canada (8):
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - CHUS-Hopital Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoledronic Acid: Zoledronic acid q 6 months plus Vitamin D and calcium supplement for 3 years in addition to concurrent radiation therapy and luteinizing hormone-releasing hormone (LHRH) therapy.
Period: Overall Study
Arm/Group | Zoledronic Acid | Control
Started | 57 | 52
Completed | 50 | 46
Not Completed | 7 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Control | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Continuous [Median (Full Range); unit: years] | 70 [51 to 87] | 71 [56 to 84] | 71 [51 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 46 | 96

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Any Bone Fracture (FABF) Rate at Three Years
Description: The time of failure was measured from the date of randomization to the date of documented bone fractures, defined as any fracture of the bone. The three-year FABF rate will be estimated by the Kaplan-Meier method.
Time Frame: From randomization to 3 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 50 | 46
percentage of participants | 98.0 [94.0 to 100.0] | 97.4 [92.3 to 100.0]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Control; The study is designed to show a 40% relative reduction in the yearly ABF hazard rate, equivalent to an improvement in a 3-year FABF rate from 88% to 92.6%. A sample size of 1030 analyzable patients with a one-sided log-rank test at α = 0.05, was calculated to provide 80% statistical power, with one interim analysis and a final analysis for efficacy using Haybittle-Peto boundaries; Test type: Superiority; p = 0.95, Log Rank

2. Secondary Outcome: Percent Change in Bone Mineral Density at 3 Years
Description: Bone mineral density (BMD) was measured by DXA scan (Dual X-ray absorptiometry) for five locations: lumbar, right total hip, left total hip, right femoral neck, and left femoral neck. The percent change at 3 years was calculated for each location by the following formula: Percent Change BMD = (BMD_3 years - BMD_Baseline)/ BMD_Baseline * 100.
Time Frame: Baseline, 3 years from start of treatment
Population: Eligible patients with baseline and 3-year BMD data at respective location
Measure: Mean (Full Range); unit: percentage of baseline value
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 50 | 46
percentage of baseline value
  Lumbar | 6 [-5 to 15] | -5 [-19 to -1]
  Hip - Right: number analyzed (Participants) | 6 | 6
  Hip - Right | -2 [-17 to 3] | -5 [-13 to 1]
  Hip - Left: number analyzed (Participants) | 19 | 9
  Hip - Left | 1 [-6 to 13] | -8 [-18 to 3]
  Femoral - Right: number analyzed (Participants) | 6 | 6
  Femoral - Right | 1 [-13 to 4] | -6 [-9 to 0]
  Femoral - Left: number analyzed (Participants) | 20 | 10
  Femoral - Left | 3 [-8 to 12] | -8 [-26 to 3]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Control; Lumbar; Test type: Superiority; p < 0.0001, t-test, 2 sided — significance level = 0.05
Statistical Analysis 2: Comparison: Zoledronic Acid vs Control; Hip - right; Test type: Superiority; p = 0.47, t-test, 2 sided — significance level = 0.05
Statistical Analysis 3: Comparison: Zoledronic Acid vs Control; Hip - left; Test type: Superiority; p = 0.0002, t-test, 2 sided — significance level = 0.05
Statistical Analysis 4: Comparison: Zoledronic Acid vs Control; Femoral - right; Test type: Superiority; p = 0.076, t-test, 2 sided — significance level = 0.05
Statistical Analysis 5: Comparison: Zoledronic Acid vs Control; Femoral - left; Test type: Superiority; p = 0.0007, t-test, 2 sided — significance level = 0.05

3. Secondary Outcome: Changes in the Functional Assessment of Cancer Therapy-General (FACT-G) at 3 Years
Description: The FACT-G is a validated, 27-item measure. In addition to a total QOL score, subscale scores for physical, functional, social and emotional well-being are produced. There are 5 responses options, with 0=Not a lot and 4=Very much. All items in a subscale are added together, multiplied by the number of items in the subscale, then divided by the number of items answered to obtain subscale totals. Scores range from 0-108 for the FACT-G total score, 0-28 for the physical, social and functional subscales, and 0-24 for the emotional subscale. Certain items, identified on the FACT-G scoring guides, must be reversed before it is added by subtracting the response from 4. All subscale totals are added together to form the FACT-G total score. Each subscale requires at least 50% of the items to be completed while the overall response rate must be greater than 80%. If items are missing, the subscale scores can be prorated. A higher score indicates better QOL.
Time Frame: Baseline, 3 years from start of treatment
Population: Eligible patients with baseline and 3-year FACT-G data
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 29 | 21
units on a scale
  Physical Subscale | -1.03 [-15 to 8] | 0.06 [-5 to 10]
  Social Subscale | -0.69 [-7.00 to 6.42] | -1.13 [-14.7 to 18.00]
  Emotional Subscale | 1.83 [-4.00 to 10.00] | 1.15 [-4.00 to 14.00]
  Functional Subscale | -1.10 [-20.8 to 5.00] | -2.76 [-11.0 to 6.00]
  Total | -1.00 [-30.7 to 19.00] | -2.77 [-27.7 to 27.00]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Control; Physical subscale; Test type: Superiority; p = 0.33, t-test, 2 sided — significance level = 0.01
Statistical Analysis 2: Comparison: Zoledronic Acid vs Control; Social subscale; Test type: Superiority; p = 0.82, t-test, 2 sided — significance level = 0.01
Statistical Analysis 3: Comparison: Zoledronic Acid vs Control; Emotional subscale; Test type: Superiority; p = 0.51, t-test, 2 sided — significance level = 0.01
Statistical Analysis 4: Comparison: Zoledronic Acid vs Control; Functional subscale; Test type: Superiority; p = 0.25, t-test, 2 sided — significance level = 0.01
Statistical Analysis 5: Comparison: Zoledronic Acid vs Control; Total; Test type: Superiority; p = 0.63, t-test, 2 sided — significance level = 0.01

4. Secondary Outcome: Utility of the Use of Bisphosphonates as Assessed by Quality-adjusted Survival
Description: The EQ-5D is a standardized instrument for measuring generic health status used to generate health utilities, used to derive quality adjusted survival. Quality adjusted survival is computed using the weighted sum of times in different health states added up to a total quality-adjusted survival time. The log-rank test is used to compare quality-adjusted survivals between the treatment arms.
Time Frame: From pre-treatment to 3 years from start of treatment
Population: Eligible patients with baseline and follow-up EQ-5D scores, resulting in only 59 patients (no deaths), less than half of enrolled patients (and less than 5% of planned enrollment), which is extremely problematic as it can lead to selection bias, especially with even fewer patients with follow-up scores. Therefore analysis was not conducted.
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Zoledronic Acid | Control
Serious Adverse Events (participants affected / at risk) | 8/50 | 5/46
Other Adverse Events (participants affected / at risk) | 45/50 | 38/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=50) | Control (N=46)
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Uveitis NOS (Eye disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 1
Colonic haemorrhage (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 0 | 1
Gait abnormal NOS (General disorders) | 0 | 1
Fracture NOS (Injury, poisoning and procedural complications) | 1 | 0
Vessel injury-artery: Carotid (Injury, poisoning and procedural complications) | 1 | 0
Lymphopenia (Investigations) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness, generalized or specific area (not due to ne (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal/genitourinary - Other: (Renal and urinary disorders) | 2 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=50) | Control (N=46)
Hemoglobin (Blood and lymphatic system disorders) | 13 | 11
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 7 | 4
Diarrhoea NOS (Gastrointestinal disorders) | 9 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 3
Gastrointestinal - Other: (Gastrointestinal disorders) | 3 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Proctitis NOS (Gastrointestinal disorders) | 3 | 5
Rectal hemorrhage (Gastrointestinal disorders) | 4 | 9
Constitutional Symptoms - Other: (General disorders) | 4 | 2
Edema: limb: (General disorders) | 7 | 2
Fatigue (General disorders) | 23 | 15
Pain - Other: (General disorders) | 5 | 1
Pain NOS (General disorders) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 4 | 1
Leukopenia NOS (Investigations) | 5 | 2
Lymphopenia (Investigations) | 7 | 5
Metabolic/laboratory - Other: (Investigations) | 5 | 2
Platelet count decreased (Investigations) | 4 | 1
Weight increased (Investigations) | 4 | 0
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal/soft tissue - Other: (Musculoskeletal and connective tissue disorders) | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Depression (Psychiatric disorders) | 6 | 3
Insomnia (Psychiatric disorders) | 3 | 2
Libido decreased (Psychiatric disorders) | 5 | 4
Pollakiuria (Renal and urinary disorders) | 20 | 13
Renal/genitourinary - Other: (Renal and urinary disorders) | 3 | 4
Urinary incontinence (Renal and urinary disorders) | 5 | 4
Urinary retention (Renal and urinary disorders) | 3 | 5
Erectile dysfunction NOS (Reproductive system and breast disorders) | 9 | 6
Gynaecomastia (Reproductive system and breast disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Hot flushes NOS (Vascular disorders) | 27 | 25

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 109 subjects accrued out of 1272 planned, less than 10% than what was planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.